CLINICAL TRIAL: NCT02820363
Title: A Prospective, Randomized Multicenter Controlled Trial of CERAMENT™|G as Part of Surgical Repair of Open Diaphyseal Tibial Fractures
Brief Title: Study Evaluating CERAMENT™|G in Open Diaphyseal Tibial Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BONESUPPORT AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN001 - FORTIFY
Record Dates: First submitted 2016-06-27; First posted 2016-07-01 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Tibial Fracture
Keywords: wound; open fracture; fracture; tibial
MeSH Terms: conditions — Tibial Fractures; Wounds and Injuries; Fractures, Open; Fractures, Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Test (Experimental): Tibial fracture fixation with IM Nail. Apply CERAMENT™|G applied to bony void(s).
  Interventions: Device: CERAMENT|G; Procedure: SOC treatment
- Control (Active Comparator): Tibial fracture fixation with IM nail.
  Interventions: Procedure: SOC treatment

INTERVENTIONS:
Device: CERAMENT|G — Surgical repair of tibia fracture, CERAMENT™|G applied to bony voids.
  Arms: Test
Procedure: SOC treatment — surgical repair of tibial fracture

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of CERAMENT™|G used in conjunction with standard-of-care treatment compared to standard-of-care treatment alone in the care of subjects with open fractures of the tibial diaphysis.

DETAILED DESCRIPTION:
CERAMENT™|G is a resorbable, gentamicin containing ceramic bone graft indicated to fill bony voids or gaps which are not intrinsic to the stability of the bony structure and where there is risk of bacterial contamination.

ELIGIBILITY:
1. Male or female 18-21 years of age with radiographic evidence on plain x-rays of proximal and distal tibial physeal closure, OR male or female 22-75 years of age
2. Gustilo-Anderson Grade II, IIIA, or IIIB open tibial shaft fracture (with or without involvement of the tibial plateau or pilon/plafond) amenable to fixation with an intramedullary nail
3. Bone loss at the fracture site must have a radiographic apparent bone gap (RABG) between 3 and 27.5 millimeters.
4. Life expectancy of at least 1 year
5. Patient is willing to provide informed consent, is geographically stable and able to comply with the required follow up visits, testing schedule and medication regimen
6. Adequate soft tissue coverage at the fracture site (through primary closure or surgical reconstruction, including local and free soft tissue transfer)
7. Definitive wound closure within 14 days of the initial injury
8. Unilateral fracture, or, in the case of individually-qualifying bilateral open tibia fractures, the more severe of the bilateral fractures.

Patients will be excluded if ANY of the following conditions apply:

1. Pregnant or breastfeeding women or planning on becoming pregnant during the investigational period
2. Patient is currently participating in an investigational drug or other device study or previously enrolled in this study
3. Renal failure or documented chronic kidney disease with serum creatinine ≥3.5 mg/L or being treated with dialysis
4. Known hypersensitivity to aminoglycoside antibiotics, calcium sulfate or calcium hydroxyapatite
5. Pre-existing calcium metabolism disorder
6. Uncontrolled diabetes mellitus (hemoglobin A1c levels > 10%)
7. A current endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, hyperthyroidism, parathyroid hormone disorder, Ehler-Danlos syndrome, osteogenesis imperfecta)
8. Neuromuscular disorders such as myasthenia gravis or Parkinson's disease
9. Currently has untreated malignant neoplasm(s), or is currently undergoing radiation therapy or chemotherapy
10. Previous history of osteomyelitis in the index limb
11. Ipsilateral tibial plateau or pilon/plafond fractures requiring a reconstruction that interferes with or prohibits the use of an intramedullary nail to stabilize the tibial shaft fracture or, in the opinion of the investigator, the treatment and/or rehabilitation of such fracture(s) would substantially interfere with the treatment, rehabilitation or other requirements of open tibial shaft fractures enrolled under this protocol.
12. Other ipsilateral lower extremity fracture(s) if, in the opinion of the investigator, the treatment and/or rehabilitation of such fracture(s) will substantially interfere with the treatment, rehabilitation or other requirements outlined in this protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Composite of absence of deep infection at fracture site, absence of secondary procedures intended to promote fracture union, and improvement in the SF-36v2 PCS. | 12 months
  Absence of secondary procedures, absence of infection.
Serious device related adverse events | 12 months
  for the test (CERAMENT™|G) arm

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R. Dirschl, MD, Principal Investigator — The University of Chicago Medicine
Locations (31):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Irvine, California
  - University of Southern California, Los Angeles, California
  - Cedars Sinai Medical Orthopedic, Los Angeles, California
  - Harbor-UCLA Medical Center, Los Angeles, California
  - Denver Health Medical Center, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - University of Missouri Health, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - New York University, Bellevue Hospital, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Department of Orthopedics Greenville Health System, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center, San Antonio, Texas
  - West Virginia University, Morgantown, West Virginia
- Germany (7):
  - Klinikum Bayreuth, Bayreuth
  - Essen University Hospital, Essen
  - BG Hospital Ludwigshafen, Ludwigshafen
  - Universitätsmedizin Mainz, Mainz
  - Rechts der Isar Hospital, Munich
  - LMU Munich, Munich
  - Universitätsklinikum Regensburg, Regensburg
- Samodzielny Publiczny Wojewodzki Szpital, Szczecin, Poland
- United Kingdom (6):
  - University Hospital Coventry, Coventry
  - The Royal London Hospital, London
  - King's College Hospital, London
  - Imperial College, London
  - University Hospitals, Manchester
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No